CLINICAL TRIAL: NCT01065935
Title: A Multicenter, Multinational, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Aerosolized ALN-RSV01 Plus Standard of Care in Lung Transplant Patients Infected With Respiratory Syncytial Virus (RSV)
Brief Title: Phase 2b Study of ALN-RSV01 in Lung Transplant Patients Infected With Respiratory Syncytial Virus (RSV)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALN-RSV01-109
Record Dates: First submitted 2010-02-05; First posted 2010-02-10 (Estimated); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: ALN-RSV01; RSV; Respiratory Syncytial Virus
MeSH Terms: conditions — Respiratory Syncytial Virus Infections | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ALN-RSV01 (Active Comparator)
  Interventions: Drug: ALN-RSV01
- Normal saline (Placebo Comparator)
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: ALN-RSV01 — Administered by nebulization once daily for 5 days
  Arms: ALN-RSV01
Drug: Normal Saline — Administered by nebulization once daily for 5 days
  Arms: Normal saline

SUMMARY:
To evaluate the efficacy and safety of ALN-RSV01 plus standard of care in RSV infected lung transplant patients

ELIGIBILITY:
Inclusion Criteria:

* Single or bilateral lung transplant recipients
* Confirmed RSV infection
* Greater than 90 days post current lung transplant
* Rejection free for a minimum of 30 days

Exclusion Criteria:

* Known viral, bacterial, or fungal respiratory co-infection at the time of RSV diagnosis
* Bronchiolitis obliterans syndrome (BOS) Grade 3 or any BOS with FEV1 that has not been stable for at least 3 months
* Use of alemtuzumab within 9 months prior to screening, anti-thymocyte globulin (ATG) within 90 days of screening or prednisone or equivalent as maintenance therapy
* Active treatment for acute graft rejection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2010-02; Primary Completion 2012-04 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
The occurrence of new or progressive BOS grade 0p through 3 in RSV-infected lung transplant recipients | 180 days after randomization

SECONDARY OUTCOMES:
Proportion of patients with FEV1 >80% of pre-infection baseline value | 90 and 180 days after randomization
RSV symptoms as measured by mean cumulative daily total symptom score | 14 days after randomization
Viral load as measured by viral area under the curve (AUC) | 6 days after randomization
All cause mortality | Throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Martin Zamora, MD, Principal Investigator — University of Colorado, Denver; Alan Glanville, MB BS MD Syd, FRACP, Principal Investigator — St. Vincents Hospital NSW W Australia; Jens T Gottlieb, MD, Principal Investigator — Hannover Medical School
Locations (31):
- United States (16):
  - Clinical Site, Phoenix, Arizona
  - Clinical Site, Los Angeles, California
  - Clinical Site, Denver, Colorado
  - Clinical Site, Tampa, Florida
  - Clinical Site, Atlanta, Georgia
  - Clinical Site, Chicago, Illinois
  - Clinical Site, Boston, Massachusetts
  - Clinical Site, Ann Arbor, Michigan
  - Clinical Site, St Louis, Missouri
  - Clinical Site, New York, New York
  - Clinical Site, Cleveland, Ohio
  - Clinical Site, Philadelphia, Pennsylvania
  - Clinical Site, Pittsburgh, Pennsylvania
  - Clinical Site, Nashville, Tennessee
  - Clinical Site, Dallas, Texas
  - Clinical Site, Houston, Texas
- Australia (4):
  - Clinical Site, Darlinghurst, New South Wales
  - Clinical Site, Adelaide, South Australia
  - Clinical Site, Melbourne, Victoria
  - Clinical Site, Perth, Western Australia
- Clinical Site, Vienna, Austria
- Canada (2):
  - Clinical Site, Edmonton, Alberta
  - Clinical Site, Toronto, Ontario
- France (2):
  - Clinical Site, Paris
  - Clinical Site, Strasbourg
- Germany (6):
  - Clinical Site, Berlin
  - Clinical Site, Essen
  - Clinical Site, Hamburg
  - Clinical Site, Hanover
  - Clinical Site, Homburg/Saar
  - Clinical Site, Leipzig